CLINICAL TRIAL: NCT00553163
Title: Hypnotherapy for Prevention of Relapse in Ulcerative Colitis: a Randomised, Single-blind, Controlled Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient numbers of patinets in the time available
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMRP proposal no IBD 0213
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2013-11

CONDITIONS: Ulcerative Colitis
Keywords: Hypnotherapy; Prevention of relapse; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gut-focussed hypnotherapy (GFH). (Active Comparator): Gut-focussed hypnotherapy (GFH).
  Interventions: Behavioral: Gut focussed hypnotherapy
- Educational sessions (Sham Comparator): Regular sessions to learn about UC from research nurse
  Interventions: Behavioral: Control educational sessions

INTERVENTIONS:
Behavioral: Gut focussed hypnotherapy — Gut focussed hypnotherapy
  Arms: Gut-focussed hypnotherapy (GFH).
Behavioral: Control educational sessions — Control educational sessions
  Arms: Educational sessions

SUMMARY:
There is increasing evidence that worsening of ulcerative colitis (UC) can be provoked by psychological stresses. When this protocol was devised, there had been no proper scientific studies to find out whether stress reduction can improve the course of UC. Hypnotherapy is a technique by which a practitioner induces a temporary trance-like state in patients: while they are in this state, the practitioner uses suggestion to induce relaxation as well as beneficial modification of the way in which the patient experiences the gut working. In previous studies in our lab, we have shown that a single 50 minute session of hypnosis can reduce special indicators of inflammation both in the blood-stream and in the lining of the lower bowel (rectum). Furthermore, in earlier work by others, hypnosis had been shown to be effective in the treatment of patients with irritable bowel syndrome, duodenal ulcer and indigestion unassociated with ulcers.

Many patients with UC need to take the immunosuppressive drug, azathioprine, in addition to a 5ASA drug, to keep their disease under control. While azathioprine is usually effective in maintaining remission of UC, it does require regular drug checks and carries the risk of possible side-effects. We undertook a study of hypnotherapy to see whether it can prevent relapse (worsening) of UC in patients who normally need to take azathioprine to keep their UC inactive. To do this, we planned to ask 66 patients who agreed to participate in the trial to stop their azathioprine. They were then to be allocated to receive either gut-focussed hypnotherapy (44 patients) or, as a control, non-emotive educational sessions (22 patients) once a month for 3 months, with intervening self-hypnosis daily in the active arm. The numbers of patients in each group who developed relapse of their UC in a year were recorded. We diagnosed relapse from patients' diaries recording diarrhoea and bleeding, and by sigmoidoscopy.

It was hoped that this clinical trial would identify a new drug-free way of reducing the chances of relapse in patients with UC.

DETAILED DESCRIPTION:
SCIENTIFIC ABSTRACT There is increasing evidence that relapse of ulcerative colitis (UC) can be provoked by psychological stress. When this study was planned, there were no proper scientific studies to find out whether stress reduction can improve the course of UC. Hypnotherapy is a technique by which a practitioner induces a temporary trance-like state in patients: while they are in this state, the practitioner uses suggestion to induce relaxation as well as beneficial modification of the way in which the patient experiences the gut working. In previous studies in our lab, we had shown that a single session of hypnosis can reduce measures of inflammation at both systemic and rectal mucosal levels. Thus, 50 min of gut-focussed hypnosis reduced serum interleukin-6 (IL6) and non-killer (NK) cell numbers in circulating blood, as well as rectal mucosal release of interleukin-13 (IL13), substance P and histamine. Furthermore, in earlier work by others, hypnosis had been shown to be effective in the treatment of patients with irritable bowel syndrome, duodenal ulcer and indigestion unassociated with ulcers.

Many patients with UC need to take the immunosuppressive, azathioprine, in addition to a 5ASA, to keep their disease in remission. While azathioprine is usually effective in maintaining remission of UC, it does require regular drug checks and carries the risk of possible side-effects. We undertook a study of hypnotherapy to see whether it could prevent relapse of UC in patients who normally need to take azathioprine to keep their UC inactive. To do this, we planned to ask 66 patients who agreed to participate in the trial to stop their azathioprine. They were then to be allocated to receive either gut-focussed hypnotherapy (44 patients) or, as a control, non-emotive educational sessions (22 patients) once a month for 3 months, with intervening self-hypnosis daily in the active arm. We then recorded relapse rates in each group at 1 year. We diagnosed relapse from patients' diaries recording the Simple Clinical Activity Index, and by Baron score >1 at sigmoidoscopy.

It was hoped that this clinical trial would identify a new drug-free way of reducing the chances of relapse in patients with UC withdrawing from treatment with azathioprine.

ELIGIBILITY:
Inclusion Criteria:

* Inactive UC
* Age 16-75 years
* Minimum 1 year on Azathioprine or Mercaptopurine.
* Simple Colitis Activity Index (SCCAI) score <3
* Baron's sigmoidoscopic score <2 .
* In remission for at least 3 months
* No change to other maintenance therapy (including 5ASA) for at least 4 months

Exclusion Criteria:

* Use of prednisolone orally or topically, or of topical 5ASA for at least 3 months Antibiotics, warfarin, anti-diarrhoeal drugs, non-steroidal anti-inflammatory drugs (NSAIDs), aspirin > 75 mg/day
* Herbal remedies
* Alcohol or drug abuse
* Pregnancy or breast feeding
* Female of child-bearing age not taking adequate contraception
* Participation in another drug trial in the previous three months
* Serious liver, renal, cardiac, respiratory, endocrine, neurological or psychiatric illness
* Already use relaxation techniques or computerized feedback

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Rampton, MAFRCP DPhil, Principal Investigator — Barts and the London/Queen Mary School of Medicine and Dentistry, London.; Anton Emmanuel, MBBS MD FRCP, Principal Investigator — University College London Hospital, London; Louise Langmead, MBBS MD MRCP, Principal Investigator — Univesity College London Hospital , London; Jeremy D Sanderson, MBBSFRCP MD, Principal Investigator — Guy's and St Thomas'NHS Trust/King's College London
Locations (3):
- United Kingdom (3):
  - Barts and The Royal London NHS Trust/Queen Mary University London/, London
  - University College Hospital London, London
  - Guy's and St Thomas' NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mawdsley JE, Rampton DS. Psychological stress in IBD: new insights into pathogenic and therapeutic implications. Gut. 2005 Oct;54(10):1481-91. doi: 10.1136/gut.2005.064261. PMID 16162953
- [Background] Bitton A, Sewitch MJ, Peppercorn MA, deB Edwardes MD, Shah S, Ransil B, Locke SE. Psychosocial determinants of relapse in ulcerative colitis: a longitudinal study. Am J Gastroenterol. 2003 Oct;98(10):2203-8. doi: 10.1111/j.1572-0241.2003.07717.x. PMID 14572569
- [Background] Levenstein S, Prantera C, Varvo V, Scribano ML, Andreoli A, Luzi C, Arca M, Berto E, Milite G, Marcheggiano A. Stress and exacerbation in ulcerative colitis: a prospective study of patients enrolled in remission. Am J Gastroenterol. 2000 May;95(5):1213-20. doi: 10.1111/j.1572-0241.2000.02012.x. PMID 10811330
- [Background] Garrett VD, Brantley PJ, Jones GN, McKnight GT. The relation between daily stress and Crohn's disease. J Behav Med. 1991 Feb;14(1):87-96. doi: 10.1007/BF00844770. PMID 2038047
- [Background] Greene BR, Blanchard EB, Wan CK. Long-term monitoring of psychosocial stress and symptomatology in inflammatory bowel disease. Behav Res Ther. 1994 Feb;32(2):217-26. doi: 10.1016/0005-7967(94)90114-7. PMID 8155059
- [Background] Mawdsley JE, Macey MG, Feakins RM, Langmead L, Rampton DS. The effect of acute psychologic stress on systemic and rectal mucosal measures of inflammation in ulcerative colitis. Gastroenterology. 2006 Aug;131(2):410-9. doi: 10.1053/j.gastro.2006.05.017. PMID 16890594
- [Background] Farhadi A, Keshavarzian A, Van de Kar LD, Jakate S, Domm A, Zhang L, Shaikh M, Banan A, Fields JZ. Heightened responses to stressors in patients with inflammatory bowel disease. Am J Gastroenterol. 2005 Aug;100(8):1796-804. doi: 10.1111/j.1572-0241.2005.50071.x. PMID 16086717
- [Background] Ewer TC, Stewart DE. Improvement in bronchial hyper-responsiveness in patients with moderate asthma after treatment with a hypnotic technique: a randomised controlled trial. Br Med J (Clin Res Ed). 1986 Nov 1;293(6555):1129-32. doi: 10.1136/bmj.293.6555.1129. PMID 3094804
- [Background] Langewitz W, Izakovic J, Wyler J, Schindler C, Kiss A, Bircher AJ. Effect of self-hypnosis on hay fever symptoms - a randomised controlled intervention study. Psychother Psychosom. 2005;74(3):165-72. doi: 10.1159/000084001. PMID 15832067
- [Background] Friedman H, Taub HA. The use of hypnosis and biofeedback procedures for essential hypertension. Int J Clin Exp Hypn. 1977 Oct;25(4):335-47. doi: 10.1080/00207147708415989. No abstract available. PMID 892940
- [Background] Horne DJ, White AE, Varigos GA. A preliminary study of psychological therapy in the management of atopic eczema. Br J Med Psychol. 1989 Sep;62(3):241-8. doi: 10.1111/j.2044-8341.1989.tb02832.x. PMID 2675960
- [Background] Shertzer CL, Lookingbill DP. Effects of relaxation therapy and hypnotizability in chronic urticaria. Arch Dermatol. 1987 Jul;123(7):913-6. PMID 3300566
- [Background] Whorwell PJ, Prior A, Faragher EB. Controlled trial of hypnotherapy in the treatment of severe refractory irritable-bowel syndrome. Lancet. 1984 Dec 1;2(8414):1232-4. doi: 10.1016/s0140-6736(84)92793-4. PMID 6150275
- [Background] Gonsalkorale WM, Houghton LA, Whorwell PJ. Hypnotherapy in irritable bowel syndrome: a large-scale audit of a clinical service with examination of factors influencing responsiveness. Am J Gastroenterol. 2002 Apr;97(4):954-61. doi: 10.1111/j.1572-0241.2002.05615.x. PMID 12003432
- [Background] Zijlstra FJ, van den Berg-de Lange I, Huygen FJ, Klein J. Anti-inflammatory actions of acupuncture. Mediators Inflamm. 2003 Apr;12(2):59-69. doi: 10.1080/0962935031000114943. PMID 12775355
- [Background] Naito A, Laidlaw TM, Henderson DC, Farahani L, Dwivedi P, Gruzelier JH. The impact of self-hypnosis and Johrei on lymphocyte subpopulations at exam time: a controlled study. Brain Res Bull. 2003 Dec 30;62(3):241-53. doi: 10.1016/j.brainresbull.2003.09.014. PMID 14698357
- [Background] Gruzelier J, Smith F, Nagy A, Henderson D. Cellular and humoral immunity, mood and exam stress: the influences of self-hypnosis and personality predictors. Int J Psychophysiol. 2001 Aug;42(1):55-71. doi: 10.1016/s0167-8760(01)00136-2. PMID 11451479
- [Background] Kiecolt-Glaser JK, Marucha PT, Atkinson C, Glaser R. Hypnosis as a modulator of cellular immune dysregulation during acute stress. J Consult Clin Psychol. 2001 Aug;69(4):674-82. doi: 10.1037//0022-006x.69.4.674. PMID 11550733
- [Background] Zachariae R, Hansen JB, Andersen M, Jinquan T, Petersen KS, Simonsen C, Zachariae C, Thestrup-Pedersen K. Changes in cellular immune function after immune specific guided imagery and relaxation in high and low hypnotizable healthy subjects. Psychother Psychosom. 1994;61(1-2):74-92. doi: 10.1159/000288872. PMID 8121979
- [Background] Wood GJ, Bughi S, Morrison J, Tanavoli S, Tanavoli S, Zadeh HH. Hypnosis, differential expression of cytokines by T-cell subsets, and the hypothalamo-pituitary-adrenal axis. Am J Clin Hypn. 2003 Jan;45(3):179-96. doi: 10.1080/00029157.2003.10403525. PMID 12570090
- [Background] Hawthorne AB, Logan RF, Hawkey CJ, Foster PN, Axon AT, Swarbrick ET, Scott BB, Lennard-Jones JE. Randomised controlled trial of azathioprine withdrawal in ulcerative colitis. BMJ. 1992 Jul 4;305(6844):20-2. doi: 10.1136/bmj.305.6844.20. PMID 1638191
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] BARON JH, CONNELL AM, LENNARD-JONES JE. VARIATION BETWEEN OBSERVERS IN DESCRIBING MUCOSAL APPEARANCES IN PROCTOCOLITIS. Br Med J. 1964 Jan 11;1(5375):89-92. doi: 10.1136/bmj.1.5375.89. No abstract available. PMID 14075156
- [Background] Gonsalkorale WM, Whorwell PJ. Hypnotherapy in the treatment of irritable bowel syndrome. Eur J Gastroenterol Hepatol. 2005 Jan;17(1):15-20. doi: 10.1097/00042737-200501000-00004. PMID 15647634
- [Background] Toomey TC, Mann JD, Abashian S, Thompson-Pope S. Relationship between perceived self-control of pain, pain description and functioning. Pain. 1991 May;45(2):129-133. doi: 10.1016/0304-3959(91)90177-Y. PMID 1876418
- [Background] Reynaert C, Janne P, Donckier J, Buysschaert M, Zdanowicz N, Lejeune D, Cassiers L. Locus of control and metabolic control. Diabete Metab. 1995 Jun;21(3):180-7. PMID 7556809
- [Background] Velayos FS, Terdiman JP, Walsh JM. Effect of 5-aminosalicylate use on colorectal cancer and dysplasia risk: a systematic review and metaanalysis of observational studies. Am J Gastroenterol. 2005 Jun;100(6):1345-53. doi: 10.1111/j.1572-0241.2005.41442.x. PMID 15929768
- [Background] Anbar RD. Self-hypnosis for the treatment of functional abdominal pain in childhood. Clin Pediatr (Phila). 2001 Aug;40(8):447-51. doi: 10.1177/000992280104000804. PMID 11516052
- [Background] Conroy SP, Mayberry JF. Patient information booklets for Asian patients with ulcerative colitis. Public Health. 2001 Nov;115(6):418-20. doi: 10.1038/sj/ph/1900799. PMID 11781853
- [Background] Maunder RG, Greenberg GR, Hunter JJ, Lancee WJ, Steinhart AH, Silverberg MS. Psychobiological subtypes of ulcerative colitis: pANCA status moderates the relationship between disease activity and psychological distress. Am J Gastroenterol. 2006 Nov;101(11):2546-51. doi: 10.1111/j.1572-0241.2006.00798.x. Epub 2006 Oct 4. PMID 17029612
- [Background] Wallston BS, Wallston KA, Kaplan GD, Maides SA. Development and validation of the health locus of control (HLC) scale. J Consult Clin Psychol. 1976 Aug;44(4):580-5. doi: 10.1037//0022-006x.44.4.580. No abstract available. PMID 939841
- [Background] Hilgard ER, Weitzenhoffer AM, Gough P. INDIVIDUAL DIFFERENCES IN SUSCEPTIBILITY TO HYPNOSIS. Proc Natl Acad Sci U S A. 1958 Dec 15;44(12):1255-9. doi: 10.1073/pnas.44.12.1255. No abstract available. PMID 16590342
- [Background] Guyatt G, Mitchell A, Irvine EJ, Singer J, Williams N, Goodacre R, Tompkins C. A new measure of health status for clinical trials in inflammatory bowel disease. Gastroenterology. 1989 Mar;96(3):804-10. PMID 2644154
- [Background] Tibble JA, Sigthorsson G, Bridger S, Fagerhol MK, Bjarnason I. Surrogate markers of intestinal inflammation are predictive of relapse in patients with inflammatory bowel disease. Gastroenterology. 2000 Jul;119(1):15-22. doi: 10.1053/gast.2000.8523. PMID 10889150
- [Background] van Toorenenbergen AW, Oranje AP. Comparison of serum tryptase and urine N-methylhistamine in patients with suspected mastocytosis. Clin Chim Acta. 2005 Sep;359(1-2):72-7. doi: 10.1016/j.cccn.2005.03.041. PMID 15913591
- [Background] Zocco MA, dal Verme LZ, Cremonini F, Piscaglia AC, Nista EC, Candelli M, Novi M, Rigante D, Cazzato IA, Ojetti V, Armuzzi A, Gasbarrini G, Gasbarrini A. Efficacy of Lactobacillus GG in maintaining remission of ulcerative colitis. Aliment Pharmacol Ther. 2006 Jun 1;23(11):1567-74. doi: 10.1111/j.1365-2036.2006.02927.x. PMID 16696804
- [Background] Bergman R, Parkes M. Systematic review: the use of mesalazine in inflammatory bowel disease. Aliment Pharmacol Ther. 2006 Apr 1;23(7):841-55. doi: 10.1111/j.1365-2036.2006.02846.x. PMID 16573787
- [Background] Shetty A, Kalantzis C, Polymeros D, Vega R, Abraham S, Forbes A. Hypnotherapy for inflammatory bowel disease- a randomised, placebo-controlled trial. Gut 2004;53:A226
- [Background] Mawdsley JE, Jenkins D, Macey MG, Rampton DS. Natural Killer cells are increased by psychological stress and decreased by hypnotherapy in ulcerative colitis. Gut 2005; 54 (Suppl II): A23
- [Background] Mawdsley JE, Jenkins D, Macey MG, Rampton DS. Hypnotherapy decreases rectal mucosal release of substance P, histamine and IL-13 in patients with active UC. Gut 2006; 55 (Suppl II): A75
- [Background] Emmanuel AV, Storrie JB, Butcher L et al. Is targeting locus of control a desirable outcome of biofeedback in functional constipation ? Gut 2007;56, suppl 11:A63.
- [Background] Rampton DS, Shanahan S. Fast facts: Inflammatory Bowel Disease. Health Press, 2nd ed, 2006.
- [Background] Mawdsley JE, Rampton DS. Serum IL-13 concentrations are raised in active ulcerative colitis and correlate with disease activity and mucosal inflammation. Gut 2005; 54 (Suppl IV): A165
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We aimed to recruit 66 patients from across London, but after >3 years could recruit only 26. Reasons for failure to complete recruitment included the relative rarity of this patient-group (ie with inactive ulcerative colitis (UC) for some years while on thiopurine, willing to stop the drug, and with time to complete the intensive programme).
Groups:
- Gut-focussed Hypnotherapy (GFH): Patients given gut-focussed hypnotherapy (GFH).after withdrawing from thiopurine
- Control Educational Sessions: Patients given control educational sessions after withdrawing from thiopurines
Period: Overall Study
Arm/Group | Gut-focussed Hypnotherapy (GFH) | Control Educational Sessions
Started | 16 | 10
Completed | 16 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with inactive UC withdrawing from thiopurines
Groups:
- Gut-focussed Hypnotherapy: 16 Patients with inactive ulcerative colitis given gut-focussed hypnotherapy
- Controlled Educational Sessions: 10 Patients with inactive ulcerative colitis given educational sessions
- Total: Total of all reporting groups
Arm/Group | Gut-focussed Hypnotherapy | Controlled Educational Sessions | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Continuous [Median (Full Range); unit: years] — Age of subjects in years, 22-65 years
  years | 31 [22 to 65] | 48 [29 to 63] | 35 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Relapse at 1 Year
Description: The number of patients suffering a relapse was compared between the two treatment groups, and was the primary outcome parameter of this study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- UC Patients Given Gut-focussed Hypnotherapy: Gut-focussed hypnotherapy (GFH). Subjects were seen at 6 face-to-face visits in the 13 week treatment period (weeks 1, 2, 3, 5, 9 and 13).
- UC Patients Given Control Educational Sessions: Controlled educational sessions:Subjects were seen at 4-weekly intervals (a total of 4 face-to-face visits in the 13 week treatment, at weeks 1, 5, 9 and 13),
Arm/Group | UC Patients Given Gut-focussed Hypnotherapy | UC Patients Given Control Educational Sessions
Number analyzed (Participants) | 16 | 10
Participants | 8 | 7

2. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) at Week 13
Description: IBDQ (standard measure of IBD patients' Quality of life (QoL) (Irvine et al 1982 approx). The IBDQ is a validated and reliable tool to measure of health-related quality of life in adult patients with IBD. The questionnaire consists of 32 questions scored in four domains: bowel symptoms, emotional health, systemic systems and social function. Scores range from 1 (poorest QoL) to 7 (best QoL). Higher scores indicate better QoL. Lowest score 7, highest score 224.
Time Frame: 13 weeks
Population: Patients all assessed at 13 weeks (end of treatment phase). 4 hypnotherapy and 1 control patient failed to complete their questionnaires
Measure: Median (Full Range); unit: units on a scale
Groups:
- UC Patients Given Gut-focussed Hypnotherapy: Gut-focussed hypnotherapy (GFH).Subjects were seen at 6 face-to-face visits in the 13 week treatment period (weeks 1, 2, 3, 5, 9 and 13).
Arm/Group | UC Patients Given Gut-focussed Hypnotherapy | UC Patients Given Control Educational Sessions
Number analyzed (Participants) | 12 | 9
units on a scale | 195 [114 to 212] | 192 [170 to 212]

3. Secondary Outcome: Hospital Anxiety and Depression Score-Anxiety, (HADSA) at Week 13
Description: Measure of anxiety, HADS Hospital anxiety and depression scale. HADS questionnaire consists of a 14 question validated questionnaire, developed to measure anxiety and depression in the hospital setting. Each item is answered by the patient on a four point (0-3) response category so the possible scores range from 0 (minimum) to 21 (maximum) for anxiety and 0 (minimum) to 21 (maximum) for depression. Higher scores indicate worse outcome,
Time Frame: 13 weeks
Population: 4 hypnotherapy and 1 control patient failed to complete their questionnaires
Measure: Median (Full Range); unit: score on a scale
Groups:
- UC Patients Given Gut-focussed Hpynotherapy: Gut-focussed hypnotherapy (GFH).Subjects were seen at 6 face-to-face visits in the 13 week treatment period (weeks 1, 2, 3, 5, 9 and 13).
Arm/Group | UC Patients Given Gut-focussed Hpynotherapy | UC Patients Given Control Educational Sessions
Number analyzed (Participants) | 12 | 9
score on a scale | 7 [3 to 11] | 10 [4 to 14]

4. Secondary Outcome: Hospital Anxiety and Depression Score-Depression (HADSD)
Description: Measure of depression. Each item is answered by the patient on a four point (0-3) response category so the possible scores range from 0 to 21 for anxiety and 0 to 21 for depression. Each item is answered by the patient on a four point (0-3) response category so the possible scores range from 0 (minimum) to 21 (maximum) for anxiety and (minimum) to 21 (maximum) for depression. Higher scores worse outcome.
Time Frame: 13 weeks
Population: 4 hypnotherapy and 1 control patient failed to complete their questionnaires
Measure: Median (Full Range); unit: units on a scale
Groups:
- UC Patients Given Gut-focussed Hypnotherapy: Gut-focussed hypnotherapy (GFH). Session one was spent familiarising the patient with the process. Subjects were seen at 6 face-to-face visits in the 13 week treatment period (weeks 1, 2, 3, 5, 9 and 13). After the end of the initial 13 week period, patients were asked to continue to practise self-hypnosis, and were phoned monthly by the therapist
- UC Patients Given Control Educational Sessions: Controlled educational sessions: Subjects were seen at 4-weekly intervals (a total of 4 face-to-face visits in the 13 week treatment, at weeks 1, 5, 9 and 13), and received a phone call at weekly intervals from the therapist to monitor progress and field questions. After the end of the initial 13 week period, patients were phoned monthly by the therapist. No attempt was made to offer any form of relaxation techniques to these patients.
Arm/Group | UC Patients Given Gut-focussed Hypnotherapy | UC Patients Given Control Educational Sessions
Number analyzed (Participants) | 12 | 9
units on a scale | 1.5 [0 to 8] | 4 [0 to 8]

5. Secondary Outcome: Perceived Stress Questionnaire-Recent (PSQ-R)
Description: Measure of recent psychological stress. THE PSQ R consists of a 30 question questionnaires: recent, in which the statements used apply to the last month in which used statements apply to the last two years (Appendix 1.3). The score for both recent and general stress levels were stated as the PSQ index ranging from 0 (non-stressed) to 0.99 (highly stressed). Higher scores indicate worse outcome.
Time Frame: 13 weeks
Population: 4 hypnotherapy and 1 control patient failed to complete their questionnaires
Measure: Median (Full Range); unit: units on a scale
Groups:
- UC Patients Given Gut-focussed Hypnotherapy: Gut-focussed hypnotherapy (GFH). Subjects were seen at 6 face-to-face visits in the 13 week treatment period (weeks 1, 2, 3, 5, 9 and 13
Arm/Group | UC Patients Given Gut-focussed Hypnotherapy | UC Patients Given Control Educational Sessions
Number analyzed (Participants) | 12 | 9
units on a scale | 0.3 [0.1 to 0.6] | 0.4 [0.1 to 0.7]

ADVERSE EVENTS:
Groups:
- Gut-focussed Hypnotherapy (GFH): Patients given gut-focussed hypnotherapy (GFH).after withdrawing from thiopurine.
  No adverse events apart from relapse
- Controlled Educational Sessions: Patients given controlled educational sessions after withdrawing from thiopurines No adverse events apart from relapse
Arm/Group | Gut-focussed Hypnotherapy (GFH) | Controlled Educational Sessions
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes